CLINICAL TRIAL: NCT02604771
Title: An Epidemiological Study to Evaluate Standard Daily Practice in Managing Patients With Arterial Hypertension
Brief Title: Egypt Hypertension Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00249
Record Dates: First submitted 2015-08-18; First posted 2015-11-13 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Different Classes of the Antihypertensive Treatment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is an epidemiological non-interventional trial that aims to evaluate standard daily practice in managing patients with arterial hypertension. The trial only records real-life clinical practice with no additional diagnostic or monitoring procedures.

The study is purposed to collect the following Egypt-specific epidemiology data on hypertension: demographic data, patients' characteristics, and patients' management/treatment in order to reach its rationale.

DETAILED DESCRIPTION:
This study is aimed to evaluate response rate of the antihypertensive treatment with Thiazide Diuretics, calcium antagonist, Angiotensin Converting enzyme Inhibitor, Angiotensin II receptor blocker, and Beta Blocker in real life practice, and to collect the following Egypt-specific epidemiology data on hypertensive patients: demographic data, patents characteristics, and patients' management/treatment.

Approximately 300 sites will be participating (1 investigator per site; 300 investigators). Patients that are to be enrolled will either be newly diagnosed with hypertension, or on current antihypertensive treatment, compiling a total of 3000 patients (21 years, or older). The study will be conducted in two sequential phases; the first phase will include 150 sites from Cairo, Giza and Alexandria aiming to reach 1500 patients followed by a second phase which will include 150 sites from Delta and Upper Egypt aiming to reach 1500 patients. Epidemiological data collection will take place at a single visit and Laboratory Investigations will be requested in the first visit. Patients will be followed for 3 visits with the investigator. The investigator will complete a Patient Record Form (PRF) with the patient's data: demographics, history, current antihypertensive drug treatment/treatment changes, results of physical examination, blood pressure (SBP/DBP), heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Males or female aged >21 years
* Subject population with newly diagnosed essential arterial hypertension
* Subject population with essential arterial hypertension currently receiving treatment with any of the following antihypertensive classes: a Thiazide Diuretics, calcium antagonist, Angiotensin Converting enzyme Inhibitor, Angiotensin II receptor blocker and Beta Blocker for at least 3 months.
* Females of childbearing potential must use a reliable method of contraception.
* Subject willing to give written informed consent

Exclusion Criteria:

* If participating in any clinical trial, the subject cannot take part in this study.
* Pregnancy and lactation.
* Patients not willing to give Informed Consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be collected from private care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2016-04-03 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
To insert number of hypertensive patients with SBP that are reaching treatment goals | 12 weeks +- 2
  To insert number of patients with Systolic Blood pressure reaching treatment goals according to the ESC 2013 criteria (Systolic blood pressure <140 mmHg* in patients) after being treated with anti-hypertensive medication/s for at least 3 months.

SECONDARY OUTCOMES:
Insert number of patients on antihypertensive pharmacological treatment reaching the DBP goals | 12 +- 2 weeks
  Inserting number of SBP patients on antihypertensive treatment reaching the DBP goals according to the Europian Society of Cardiology (ESC) 2013 guidelines.
Insert number of patients on antihypertensive pharmacological treatment reaching SBP goals | 12 +- 2 weeks
  Inserting number of patients on antihypertensive treatment reaching combined SBP &DBP treatment goals according to Europian Society of Cardiology (ESC) 2013 guidelines.
Insert epidemiological information on antihypertensive patients in study | 12 +- 2 weeks
  * Documenting epidemiological data from the Hypertensive patients during the visit via the investigator asking them and documenting it (Age)
  * Documenting any associated major cardiovascular co-morbid diseases by the investigator asking the patient or checking patient history then writing it down in Case Report Form (CRF).
Insert treatment & managing plan of antihypertensive pharmacological treatment | 12 +- 2 weeks
  * Investigator is to document the treatment/management with any changes in it chosen for the patient.
  * to document tolerability via questionnaire.
Insert number of patients on antihypertensive pharmacological treatment reaching DBP goals | 12+- 2 weeks
  Inserting number of patients on antihypertensive treatment reaching combined SBP &DBP treatment goals according to Europian Society of Cardiology (ESC) 2013 guidelines
Insert epidemiological information on antihypertensive patients in study | 12 +- 2 weeks
  * Documenting epidemiological data from the Hypertensive patients during the visit via the investigator asking them and documenting it (Weight)
  * Documenting any associated major cardiovascular co-morbid diseases by the investigator asking the patient or checking patient history then writing it down in Case Report Form (CRF).
Insert epidemiological information on antihypertensive patients in study | 12 +- 2 weeks
  * Documenting epidemiological data from the Hypertensive patients during the visit via the investigator asking them and documenting it (gender)
  * Documenting any associated major cardiovascular co-morbid diseases by the investigator asking the patient or checking patient history then writing it down in Case Report Form (CRF).
Insert treatment & managing plan of antihypertensive pharmacological treatment | 12 +- 2 weeks
  * Investigator is to document the treatment/management with any changes in it chosen for the patient.
  * to document stability of the patient in the Case report form (CRF).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Saleh, PHD, Principal Investigator — Proffessor Cardiology Ain Shams University; Mohamed Mohsen Ibrahim, PHD, Principal Investigator — Cairo University; Mohamed Awad Taher, PHD, Principal Investigator — Ain Shams University; Khaled Leon, PHD, Principal Investigator — National Heart Institute; Ahmed Shawky, PHD, Principal Investigator — Ain Shams University
Locations (1):
- Research Site, Egypt, Cairo Governorate, Egypt

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3936&filename=1_NIS_D1843R00249_CSR14Feb2019%20_ready%20dor%20posting.pdf